CLINICAL TRIAL: NCT05566938
Title: Study to Design a Tailored Precision Nutrition Strategy Based on Metabotypes in the Elderly
Brief Title: Study to Design a Precision Nutrition Strategy At a Group Level in the Elderly
Acronym: NUTRIMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Consorci Sanitari del Maresme (CsdM) (Unknown); Centro de investigación biomédica en red enfermedades hepáticas y digestivas (Ciberhd) (Unknown); Bana Hosting (Unknown); Sixtemia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NUTRIMET
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Aging
Keywords: metabotypes; clusters; tailored nutrition; mhealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tailored nutritional recommendations for each metabotype (Other): Volunteers that will be clustered into metabotypes and will recieve tailored nutritional recommendations according to their metabotype.
  Interventions: Other: Tailored nutritional recommendations for each metabotype

INTERVENTIONS:
Other: Tailored nutritional recommendations for each metabotype — Tailored nutritional recommendations for each metabotype detected (at the group level), that will be delivered through a mobile application. Moreover, each volunteer will recieve individualized nutritional recommendations.

SUMMARY:
From a public health point of view, personalized nutritional recommendations, at the individual level, are difficult to achieve in the short-medium term, especially in population segments with less purchasing power. Therefore, a more realistic vision in the short term and with a more favourable cost/effectiveness ratio consists of carrying out dietary advice at the group level through the identification of metabotypes, which can be defined as groups of individuals with similar metabolic profiles. The application of tailored precision nutrition aimed at the elderly is detected as a strategy to understand the different alterations associated to aging and to design innovative nutritional interventions that address this physiological process, favouring a healthy ageing.

DETAILED DESCRIPTION:
The main objective of this study is to design a precision nutrition strategy at the group level in older people, based on the identification of metabotypes and enterotypes, and combining complementary variables such as anthropometric, biochemical and clinical biomarkers.

The specific objectives of the study are:

1. To identify metabotypes (clusters) in a cohort of older people, through an integrated approach of metabolomics, intestinal microbiota and anthropometric, biochemical and clinical biomarkers.
2. To develop digital tools, integrated into a mobile application, that allow the precise assignment of automated nutritional recommendations at the group level based on the metabotypes obtained, as well as promoting the adoption of new dietary habits through diet self-monitoring.
3. To evaluate the concordance of the nutritional recommendations generated at the group level by means of an automated system with the recommendations elaborated at the individual level by a nutritionist.

A total of 150 elderly people (age> 65 years) will be recruited. In order to identify the metabotypes, blood, urine and feces will be collected to determine biomarkers of inflammation, glucose metabolism, lipid metabolism, oxidative stress, bone health, sarcopenia, clinical biomarkers, intestinal microbiota and metabolomics. In addition, the following measures will be analyzed: food intake (3-day dietary records), anthropometric variables, blood pressure, bowel movement and stool consistency, diagnosis of dysphagia and sarcopenia, and measurement of frailty, muscle strength and physical performance. By using clustering tools, groups with similar metabolism and microbiota profiles (metabotypes and enterotypes) will be defined and the variables that contribute most significantly to the differentiation between clusters will be determined. The nutritionist team will elaborate tailored dietary advice for each cluster.

In parallel, mobile health tools will be developed in order to allow the volunteers to recieve and check these nutritional recommendations, and to facilitate behaviour change through dietary self-monitoring.

The volunteers will also recieve personalized nutritional recommendations individually. The tailored nutritional recommendations given at the group level (metabotypes) will be compared with the individually personalized recommendations. The objective is to obtain a high coincidence (> 80%) in the dietary recommendations between these two approaches.

The total duration of the study for each volunteer will be 14 months. During this period, participants will make 4 visits:

* A pre-selection visit (to check inclusion/exclusion criteria) (V0; day 1) and, if the inclusion criteria are met,
* A study visit (V1; day 5) in which samples will be collected from faeces, urine and blood; and the following will be measured: food intake (3-day dietary record), anthropometry, body composition, blood pressure, frailty, muscle strength, physical performance, bowel movement and stool consistency, diagnosis of dysphagia and sarcopenia.
* A study visit (V2; day 30) in which individualized nutritional recommendations will be provided to the volunteer by the nutritionist.
* A telephonic study visit (V3; month 14) in which an explanation of the instructions to download and run the App through the volunteer will have access to targeted dietary recommendations (according to the assigned cluster) will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 65 years of age
2. Have or have access (caregiver, family member) to a smartphone or tablet with Android operating system version 6 (API 23) or higher, with internet access
3. Have the signed informed consent before the initial screening visit

Exclusion Criteria:

1. Have food allergies or intolerances
2. Have diarrhea
3. People with irritable bowel syndrome or inflammatory bowel disease.
4. Present some severe chronic pathology with clinical manifestations such as cardiovascular disease, coronary disease, chronic kidney disease or cancer.
5. Participate or have participated in another clinical study or nutritional intervention in the 30 days prior to inclusion in the study.
6. Following a prescribed diet for any reason, including weight loss, in the past month.
7. Recent use of antibiotics in the last two weeks.
8. Consumption of prebiotics and/or probiotics in the 30 days prior to the study
9. Have a BMI <18.5 kg/m2
10. Smoke more than 10 cigarettes a day
11. Consume more than 14 standard drinking units (SDUs) of alcoholic beverages per week

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Concordance between the nutritional recommendations generated at the group level and at the individual level | At the final point (month 14)
  To assess the concordance between the two methods used (group vs individual nutritional recommendations) the following will be considered:
  * How many of the nutrients identified as main objectives match between the 2 methods (in percentage)
  * How many nutritional recommendations generated by the 2 methods agree with each other (in percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, MD, PhD, Principal Investigator — Consorci Sanitari del Maresme (CsdM)
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Spain